CLINICAL TRIAL: NCT00415051
Title: Safety and Immunogenicity of Live-Attenuated MP-12 Rift Valley Fever Vaccine in Humans, and Genetic Characterization of Virus Isolates Recovered From the Blood of Vaccinated Volunteers: A Phase II Study
Brief Title: Safety/Immunogenicity/Genetic Drift of MP-12 Rift Valley Fever Vaccine
Acronym: MP-12
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FY04-33, Log A-13698
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Results first posted 2017-02-01 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Rift Valley Fever
Keywords: Rift Valley Fever, vaccine
MeSH Terms: conditions — Rift Valley Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Group Assignment (Experimental): RVF MP-12
  Interventions: Biological: RVF MP-12

INTERVENTIONS:
Biological: RVF MP-12 — Administer 1 ml SQ

SUMMARY:
This study is to determine if a vaccine for Rift Valley Fever (RVF) is safe to give to humans. The study will examine how well the vaccine (RVF MP-12) stimulates the body's immune response (which fights off infection) and if the vaccine is stable or if the virus used to make the vaccine changes into a different form once injected into the body. Twenty healthy volunteers (18-50 years old) will be vaccinated with a single dose of undiluted RVF MP-12, injected into a muscle.

DETAILED DESCRIPTION:
Rift Valley Fever (RVF) is a mosquito-borne disease in Africa that affects both humans and animals. The disease poses a significant endemic disease threat, and the etiologic agent (RVF virus) possesses physical and biochemical characteristics that have resulted in its classification as a Category A Agent. Historically, this disease was confined to Africa. In September 2000, however, RVF appeared in the western part of the Kingdom of Saudi Arabia (843 cases with 114 deaths) and in Yemen (1,087 suspected cases with 121 deaths). It is thought that Rift Valley fever was introduced into this new geographic area through importation of infected livestock from Djibouti. Mosquito transmission has been subsequently demonstrated in these areas, suggesting that the disease may have become permanently established. A safe and effective RVF vaccine capable of inducing protective immunity after a single injection is urgently needed. Currently, no drug is available that will alter the course of the disease in humans or animals, nor is any licensed vaccine for RVF approved for human use. This protocol is an open-label, Phase II study to assess the safety, immunogenicity and genetic stability of RVF MP-12 vaccine in humans. The objectives of this study are to collect safety and immunogenicity data for an intramuscular (IM) injection of live, attenuated, mutagenized RVF 12th mutagenesis passage (MP-12) vaccine and characterize isolates of the Rift Valley fever (RVF) MP-12 vaccine recovered from blood of vaccinated volunteers using in vitro systems to evaluate genetic stability. A total of 20 volunteers will be recruited from among military and civilian persons at and around USAMRIID and from the general population in and around Frederick, Maryland, who expect to remain in the area for the duration of the study. Volunteers will be vaccinated with undiluted RVF MP-12 vaccine. Safety will be evaluated by recording the frequency and severity of clinical reactions to the vaccine, as well as by measuring complete blood counts and selected serum biochemistry (enzyme) values. Immunogenicity will be evaluated by measuring 80% plaque reduction neutralization (PRNT80) antibodies to RVF virus for periods up to 1 year following vaccination. Genetic stability of the vaccine will be evaluated by examining isolates recovered from blood of vaccinated volunteers by molecular sequencing techniques, and comparing these findings with those from the vaccine virus inoculum. Subjects will participate in the study for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 50 years old
* Free of chronic medical conditions requiring ongoing therapy and in general good health as determined by a physician investigator
* Have a current (within 30 days of scheduled blood donation for this study) complete blood (cell) count (CBC) to include a Hct and Hgb that show no evidence of anemia, and total white blood cell with differential platelet counts that are within normal range, as well as hepatic enzyme (AST, ALT, LDH) values that are within normal laboratory ranges
* Negative human immunodeficiency virus (HIV) antibody test within 3 months preceding vaccination
* No evidence of pre-existing liver disease or current infection with Hepatitis A, B, or C virus as determined by serology
* No evidence for pre-existing eye disease, as determined by fundoscopic/slit lamp examination by the study ophthalmologist other than refractory changes
* No evidence by history or serologic testing for previous infection with RVF virus or RVF vaccine
* Subjects must agree to refrain from intimate contact (sexual activity), or use barrier contraception (e.g., condoms), for the 2-week period following vaccination
* Females of child-bearing potential must have a negative serum pregnancy test on screening and the morning of vaccination prior to receipt of the vaccine and must agree to use a highly effective method of birth control during the first 3 months following receipt of the MP-12 vaccine. A highly effective method of birth control is defined as one with a failure rate of less than 1% per year. Acceptable birth control methods that meet this criterion include hormonal implants and injectables (Norplant, Dep-Provera, Lunelle, and Etonogestrel); combined oral contraceptives; the intrauterine devices (IUDs) Copper T (380-A) or Mirena (Levonorgestrel Intrauterine System); female sterilization (tubal ligation); sexual abstinence; or a vasectomized partner.
* Subjects must be medically cleared for participation by an investigator
* Subjects must expect to remain in the area for the duration of the study
* Volunteer must sign an approved informed consent
* Volunteer must be willing to return for all follow-up visits including a post-vaccination ophthalmologic visit
* Volunteer must be willing to refrain from excessive (more than individual's normal routine) exercise for a period of at least 2 weeks prior to and following vaccination
* Volunteer must be willing to abstain from drinking alcoholic beverages for a period of at least 2 weeks prior to and following vaccination. Volunteer must not be a "weekend" drinker or normally drink more than 2 drinks a day if male or 1 drink a day if female.
* Volunteer must agree to report any adverse event (AE) that may or may not be associated with administration of the test article during their participation in the study.

Exclusion Criteria:

* History or evidence of liver disease/abnormality
* History of pre-existing thymic disease or thymic dysfunction (any cellular immune or antibody disorders)
* Be taking any medication, prescription or non-prescription (excluding dietary supplements), on a regular basis with the exception of contraceptive pills. This includes the regular use of statins, non-steroidal anti-inflammatory drugs (NSAIDs), immunosuppressive agents, antivirals, topical steroidal creams, and nasal sprays. Conditions requiring intermittent medications and other decisions regarding eligibility due to medication use will be deferred to physician investigators.
* Elevation above the upper limit of laboratory normal values in liver enzymes, or history of unexplained elevation in liver enzymes
* History or evidence of eye disease (excluding changes in refraction and strabismus)
* Abnormal clinical lab results indicating evidence of anemia, immunosuppression, or immune deficiency disease
* Have donated 1 unit (500 cc) or more of blood for any reason during the 2 months (56 days) preceding administration of the vaccine (as assessed by query)
* Plan to donate blood within 1 year following receipt of the vaccine
* History or evidence of previous infection with RVF or vaccination against RVF
* Any known allergies to components of the vaccine: Human serum albumin (stabilizer), Sol-U-Pro, Neomycin (antibiotic), sorbitol, L-proline, L-arginine, monosodium glutamate (MSG), or Urea
* Administration of another vaccine within 4 weeks of RVF MP-12 vaccination
* "Weekend" drinkers, males who drink more than 2 drinks a day and females who drink more than 1 drink a day, will be excluded
* Individuals who plan to start a new exercise program within two weeks of vaccination (either two weeks prior to or two weeks following vaccination) will be excluded. Individuals who are already on a regular exercise program and who have normal transaminase levels will not be excluded but will be advised not to increase their level of activity for a period of one month (for two weeks prior to until two weeks after vaccination). Individuals who do not exercise regularly and who participate in this study will be advised not to embark on an exercise program for the same time period.
* Volunteers will be cautioned against salivary contact and contact with infants, children under the age of 8 years, adults over the age of 64 years, and anyone who is immunocompromised or in poor health. Volunteers who feel unable to comply with these restrictions will be excluded from the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2006-08; Primary Completion 2008-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Pittman, MD, Principal Investigator — USAMRIID Medical Division
Locations (1):
- US Army Medical Research Institute of Infectious Diseases, Fort Deterick, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty subjects were planned; 31 were screened, 11 did not meet the inclusion/exclusion criteria, 20 satisfied inclusion/exclusion criteria, 20 were enrolled, 1 was excluded (received another vaccine within 30 days of intended MP-12 vaccination), and 19 received vaccine and completed the study.
Period: Overall Study
Arm/Group | Single Group Assignment
Started | 20
Completed | 19
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Group Assignment
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 33 [23 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Safety as Measured by the Number of Adverse Events
Description: AE's will be assessed through study completion. Safety will be evaluated by recording the frequency of clinical reactions to the vaccine and by measuring complete blood counts and selected serum biochemistry (enzyme) values, rates of hospitalizations, and rates of lost duty/work time overall and by gender.
Time Frame: up to 1 year
Measure: Number; unit: AEs
Arm/Group | Single Group Assignment
Number analyzed (Participants) | 19
AEs
  Local AEs Related and Not Related to Study Drug | 22
  Systemic AEs Related and Not Related to Study Drug | 130

2. Secondary Outcome: Immune Response Assessed by Measuring Days to Peak Response for PRNT80 Antibodies to RVF Virus
Description: Immune response will be assessed by measuring days to peak response for PRNT80 antibodies to RVF virus
Time Frame: Days 0, 1, 2, 3, 7, 10, 14 and 28, Months 3, 6 and 12
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Single Group Assignment
Number analyzed (Participants) | 19
Days
  Days to peak PRNT80 | 71.1 (74.4)
  Days to peak PRNT80 response | 16.6 (6.7)

3. Secondary Outcome: Immune Response Assessed by Measuring Days to Peak Response for (PRNT50) RVP MP-12 Vaccine
Description: Immune response will be assessed by measuring days to peak response for PRNT50 antibodies to RVF virus
Time Frame: Days 0, 1, 2, 3, 7, 10, 14 and 28, Months 3, 6 and 12
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Single Group Assignment
Number analyzed (Participants) | 19
Days
  Days to peak PRNT50 | 82.2 (101.1)
  Days to peak PRNT50 response | 15.0 (6.8)

4. Secondary Outcome: Genetic Stability - Characterize Viral Isolate (Plasma) Frequency
Description: In vitro systems will be used to evaluate genetic stability (examining viremia levels in plasma by direct plaque assay techniques or by blind passage of plasma on Vero cells and sequencing the ribonucleic acid (RNA) and comparing these findings with those from the vaccine virus inoculum).
Time Frame: Days 0-14
Population: 1 subject was excluded for receiving another vaccination within 30 days of intended MP-12 vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Group Assignment
Number analyzed (Participants) | 19
Participants
  Day 0 after vaccination - Negative | 18
  Day 0 after vaccination - Positive | 0
  Day 1 after vaccination - Negative | 19
  Day 1 after vaccination - Positive | 0
  Day 2 after vaccination - Negative | 19
  Day 2 after vaccination - Positive | 0
  Day 3 after vaccination - Negative | 19
  Day 3 after vaccination - Positive | 0
  Day 4 after vaccination - Negative | 18
  Day 4 after vaccination - Positive | 1
  Day 5 after vaccination - Negative | 17
  Day 5 after vaccination - Positive | 2
  Day 6 after vaccination - Negative | 17
  Day 6 after vaccination - Positive | 2
  Day 7 after vaccination - Negative | 18
  Day 7 after vaccination - Positive | 1
  Day 8 after vaccination - Negative | 18
  Day 8 after vaccination - Positive | 1
  Day 9 after vaccination - Negative | 17
  Day 9 afterr vaccination - Positive | 2
  Day 10 after vaccination - Negative | 19
  Day 10 after vaccination - Positive | 0
  Day 11 after vaccination - Negative | 19
  Day 11 after vaccination - Positive | 0
  Day 12 afterr vaccination - Negative | 19
  Day 12 after vaccination - Positive | 0
  Day 13 after vaccination - Negative | 19
  Day 13 after vaccination - Positive | 0
  Day 14 after vaccination - Negative | 19
  Day 14 after vaccination - Positive | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Within 30 days post vaccination, 119 AEs (22 local and 97 systemic) were reported. Between 31 days and 1 year post vaccination, 33 systemic AEs (no local AEs) were reported. A total of 152 AEs (22 local and 130 systemic) were reported during the study.
Arm/Group | Single Group Assignment
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 19/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Group Assignment (N=19)
Headache (Nervous system disorders) | 16 (16) — < 30 Days Post Vaccination
Fatigue (General disorders) | 10 (10) — < 30 Days Post Vaccination
Flu-like symptoms (Respiratory, thoracic and mediastinal disorders) | 6 (6) — < 30 Days Post Vaccination
Fever (General disorders) | 4 (4) — < 30 Days Post Vaccination
Chills (Musculoskeletal and connective tissue disorders) | 2 (2) — < 30 Days Post Vaccination
Menstrual cramps (Reproductive system and breast disorders) | 1 (1) — < 30 Days Post Vaccination
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (6) — < 30 Days Post Vaccination
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 5 (5) — < 30 Days Post Vaccination
Sore throat (Gastrointestinal disorders) | 3 (3) — < 30 Days Post Vaccination
Blurred vision (Nervous system disorders) | 2 (2) — < 30 Days Post Vaccination
Conjunctivitis (OS) (Infections and infestations) | 1 (1) — < 30 Days Post Vaccination
Ear discomfort (Ear and labyrinth disorders) | 1 (1) — < 30 Days Post Vaccination
Throat scratchy and sore (Gastrointestinal disorders) | 1 (1) — < 30 Days Post Vaccination
Left eye itching (Eye disorders) | 1 (1) — < 30 Days Post Vaccination
Eyelid twitching (Nervous system disorders) | 1 (1) — < 30 Days Post Vaccination
Nausea (Gastrointestinal disorders) | 5 (5) — < 30 Days Post Vaccination
Diarrhea (Gastrointestinal disorders) | 4 (4) — < 30 Days Post Vaccination
Vomiting (Gastrointestinal disorders) | 2 (2) — < 30 Days Post Vaccination
Abdominal cramping (Gastrointestinal disorders) | 1 (1) — < 30 Days Post Vaccination
Dehydration (Gastrointestinal disorders) | 1 (1) — < 30 Days Post Vaccination
Cervial nodes slightly tender (Blood and lymphatic system disorders) | 1 (1) — < 30 Days Post Vaccination
Increase in bleeding post venipuncture (Blood and lymphatic system disorders) | 1 (1) — < 30 Days Post Vaccination
Muscle pain (Musculoskeletal and connective tissue disorders) | 6 (6) — < 30 Days Post Vaccination
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — < 30 Days Post Vaccination
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) — < 30 Days Post Vaccination
Lower back discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) — < 30 Days Post Vaccination
Knee joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) — < 30 Days Post Vaccination
Dental pain (Musculoskeletal and connective tissue disorders) | 1 (1) — < 30 Days Post Vaccination
Ankel pain (Musculoskeletal and connective tissue disorders) | 1 (1) — < 30 Days Post Vaccination
Stiff neck (Musculoskeletal and connective tissue disorders) | 1 (1) — < 30 Days Post Vaccination
Dizziness (Nervous system disorders) | 1 (1) — < 30 Days Post Vaccination
Lightheaded (Nervous system disorders) | 1 (1) — < 30 Days Post Vaccination
Spacey (Nervous system disorders) | 1 (1) — < 30 Days Post Vaccination
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) — < 30 Days Post Vaccination
Chest congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — < 30 Days Post Vaccination
Tenderness (vaccine site) (Skin and subcutaneous tissue disorders) | 9 (9) — < 30 Days Post Vaccination
Induration (Skin and subcutaneous tissue disorders) | 3 (3) — < 30 Days Post Vaccination
Redness (vaccine site) (Skin and subcutaneous tissue disorders) | 3 (3) — < 30 Days Post Vaccination
Clammy skin (hands) (Skin and subcutaneous tissue disorders) | 2 (2) — < 30 Days Post Vaccination
Bruise (Skin and subcutaneous tissue disorders) | 2 (2) — < 30 Days Post Vaccination
Itching (Skin and subcutaneous tissue disorders) | 2 (2) — < 30 Days Post Vaccination
Injection site warm (Skin and subcutaneous tissue disorders) | 1 (1) — < 30 Days Post Vaccination
Redness (phlebotomy site) (Skin and subcutaneous tissue disorders) | 1 (1) — < 30 Days Post Vaccination
Cold sore (Skin and subcutaneous tissue disorders) | 1 (1) — < 30 Days Post Vaccination
Allergic reaction (Immune system disorders) | 1 (1) — 31 days - 1 year post vaccine
Insomnia (Psychiatric disorders) | 1 (1) — 31 days - 1 year post vaccine
Pain (testicle) (Reproductive system and breast disorders) | 1 (1) — 31 days - 1 year post vaccine
Heart palpitations (Cardiac disorders) | 1 (1) — 31 days - 1 year post vaccine
Cold (Respiratory, thoracic and mediastinal disorders) | 2 (2) — 31 days - 1 year post vaccine
Eye twitching (Nervous system disorders) | 1 (1) — 31 days - 1 year post vaccine
Laryngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — 31 days - 1 year post vaccine
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — 31 days - 1 year post vaccine
Sore throat (Gastrointestinal disorders) | 2 (2) — 31 days - 1 year post vaccine
Emesis (Gastrointestinal disorders) | 1 (1) — 31 days - 1 year post vaccine
Indigestion (Gastrointestinal disorders) | 1 (1) — 31 days - 1 year post vaccine
Nausea (Gastrointestinal disorders) | 1 (1) — 31 days - 1 year post vaccine
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1) — 31 days - 1 year post vaccine
Muscle ache (Musculoskeletal and connective tissue disorders) | 3 (3) — 31 days - 1 year post vaccine
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — 31 days - 1 year post vaccine
Pain (chest and back) (Musculoskeletal and connective tissue disorders) | 1 (1) — 31 days - 1 year post vaccine
Pain (lower back) (Musculoskeletal and connective tissue disorders) | 1 (1) — 31 days - 1 year post vaccine
Pain (shoulder) (Musculoskeletal and connective tissue disorders) | 1 (1) — 31 days - 1 year post vaccine
Scar reconstruction ABD wall liposuction (Surgical and medical procedures) | 1 (1) — 31 days - 1 year post vaccine
Shin splints (Musculoskeletal and connective tissue disorders) | 1 (1) — 31 days - 1 year post vaccine
Shoulder injury (Injury, poisoning and procedural complications) | 1 (1) — 31 days - 1 year post vaccine
Stiff neck (Musculoskeletal and connective tissue disorders) | 1 (1) — 31 days - 1 year post vaccine
Traumatic injury to L middle finger (Injury, poisoning and procedural complications) | 1 (1) — 31 days - 1 year post vaccine
Dizziness (Nervous system disorders) | 1 (1) — 31 days - 1 year post vaccine
Migrane (Nervous system disorders) | 2 (2) — 31 days - 1 year post vaccine
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) — 31 days - 1 year post vaccine
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — 31 days - 1 year post vaccine

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No